CLINICAL TRIAL: NCT06857162
Title: Comparison of Maternal Hemodynamics During Spinal Anesthesia with Different Cesarean Delivery Positioning
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Collaborators: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Yousef Mohamed, Resident of Anethesia and Intensive Care, Aswan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 966/9/24
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-08

CONDITIONS: This Study Aims to Provide Evidence on Which Positioning Strategy Offers the Best Hemodynamic Outcomes; Maternal Hemodynamic; Maternal Positioning During CS

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (N=72): Immediate Supine Position (Active Comparator)
  Interventions: Behavioral: Positioninng during Cs
- Group В (N=72): Sitting Position (Experimental)
  Interventions: Behavioral: Positioninng during Cs
- Group С (N=72): Semi-Sitting Position (Experimental)
  Interventions: Behavioral: Positioninng during Cs

INTERVENTIONS:
Behavioral: Positioninng during Cs — 1. Group A (N=72): Immediate Supine Position (Control):
     Immediately after administering spinal anesthesia, participants will be placed in a supine position. To reduce the risk of aortocaval compression, a slight left lateral tilt (approximately 15 degrees) will be applied. This is the traditional positioning method and serves as the control group for comparison.
  2. Group В (N=72): Sitting Position:
     After spinal anesthesia, participants will be positioned in a sitting position with the ack supported at a 90-degree angle for the first 2 minutes. Knees will be bent, and feet will be supported.
  3. Group С (N=72): Semi-Sitting Position:
  After spinal anesthesia, participants will be positioned in a semi-sitting position with the back supported at the back supported at for the first 2 minutes.
  Similar to the sitting position, knees and feet will be flat.

SUMMARY:
Cesarean delivery is a common surgical procedure, and maintaining maternal hemodynamic stability during the procedure is crucial for both maternal and fetal outcomes . Hemodynamic instability, such as hypotension following spinal anesthesia, is a frequent complication and can lead to adverse maternal and neonatal outcomes. Traditionally, after spinal anesthesia, women are positioned supine, sometimes with a slight left lateral tilt to mitigate the risk of aortocaval compression . However, recent studies and clinical observations suggest that delayed supine positioning-keeping the patient in a sitting or semi-sitting position for a period following spinal anesthesiamay improve hemodynamic stability. These alternative positions may help to mitigate the abrupt drop in blood pressure commonly seen after spinal anesthesia by allowing for a more gradual redistribution of blood volume . Understanding the optimal positioning strategy could lead to improved clinical protocols that enhance maternal and fetal safety. By comparing immediate supine positioning with delayed supine positioning (in sitting and semi-sitting positions), this study aims to provide evidence on which positioning strategy offers the best hemodynamic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women scheduled for elective cesarean delivery.
* Age between 18 and 40 years.
* ASA (American Society of Anesthesiologists) physical status II.

Exclusion Criteria:

* Emergency cesarean delivery.
* Pre-existing cardiovascular disease.
* Severe preeclampsia or eclampsia.
* Multiple pregnancies.
* Known fetal anomalies.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 216 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
To compare the incidence and severity of hypotension in immediate supine, sitting, and semi-sitting positions during cesarean delivery. | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Mohamadi Eldemrdash, MD Of Anesthesia, Study Chair — Aswan University
Locations (1):
- Aswan University Hospital, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided